CLINICAL TRIAL: NCT03926546
Title: Individual Versus Group Exposure and Response Prevention Therapy for the Treatment of Obsessive-Compulsive Disorder
Brief Title: Individual Versus Group Exposure With Response Prevention (ERP) for the Treatment of Obsessive Compulsive Disorder (OCD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The former principal investigator left the institution.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric Alan Storch, Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H-44611
Record Dates: First submitted 2019-01-09; First posted 2019-04-24 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: OCD
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual ERP (Experimental): Individual Exposure and Response Prevention for OCD
  Interventions: Behavioral: ERP for Individuals
- Group ERP (Experimental): Group Exposure and Response Prevention for OCD
  Interventions: Behavioral: ERP for Individuals

INTERVENTIONS:
Behavioral: ERP for Individuals — Comparing Group vs. Individual ERP for OCD
  Other Names: ERP for Groups

SUMMARY:
The primary objective is to examine the efficacy of implementing evidence based Exposure and Response Prevention (ERP) within group therapy versus individual therapy by monitoring reduction of Obsessive-Compulsive Disorder (OCD) symptomology.

DETAILED DESCRIPTION:
The purpose of the following study is to observe the effectiveness of group Exposure and Response Prevention verses individual Exposure and Response Prevention on patients with OCD for the use of future publications.

A total of 70 individuals will be recruited through different methods. The primary recruitment sources will be through BCM Psychiatric Clinic patient flow. Although it is anticipated that most of the study recruitment will occur through normal BCM Psychiatric Clinic patient flow, study advertisements will also be circulated through several relevant sources (e.g. BCM OCD Program website, Peace of Mind Foundation website and listserv, social media pages and OCD organizations and groups). The investigators will also contact clinicians and professionals working with OCD patients (e.g., private clinics, community organizations) in the community to distribute advertisement flyers to potential participants.

Enrollment will occur in person at Baylor College of Medicine after obtaining informed consent.

Pertinent clinical information will be collected from paper or electronic medical records. Demographics (race, ethnicity, gender, education, employment status), and health history (concomitant medical history) will be collected and entered in the database. Data entered in the database will be coded. Patient identifying information such as name, address, telephone, date of birth, and medical record number will be extracted from the medical record. A study ID will be assigned to each subject. The code linking the consented subjects' clinical information to their study ID will be stored in a password protected database. The code linking key containing patient identifying information will be kept separately from the database. Any relevant paperwork, including videos, will be stored in a locked file cabinet in the PIs office.

Prospective data collection will continue for those subjects that consent to participate in the study.

Investigators wishing to utilize the information collected in this database must show proof of an IRB approved protocol that will be reviewed by the PI of this database registry before information can be released. Depending on the purpose of the research, data will be shared without identifiers if possible. If requested, data can be sent coded to the investigator. Only those subjects that fit inclusion criteria for the proposed research and specify that they consent to be contacted about other research will be shared with the other requesting investigators. Other investigators will not have access to the document that links coded data to identifiers.

Participants will be randomly assigned (1:1) to receive either individual therapy (i.e., 12 individual ERP sessions, each 45-60 minutes, offered twice weekly for a total of six weeks) or group therapy (a total of 6 group ERP sessions, each 120 minutes, offered weekly for 6 weeks). Sessions will be led by an ERP trained mental health professional or trainee under the supervision of a licensed mental health professional. Both the individual and group participants will receive a total of 12 hours of ERP over the span of six weeks. However, those assigned to group therapy will meet for 2 hours weekly versus those assigned to individual therapy will meet for 1 hour twice weekly. Each session will consist of completed measures and therapy involving ERP for the entirety of the six weeks. Participants assigned to the group therapy protocol will be placed in groups, each consisting of 5-8 individuals, with two therapists per group.

In the groups, Session 1 will focus on psychoeducation about ERP and OCD. Sessions 2-5 will involve ERP tasks. Session 6 will focus on relapse prevention strategies. In individual treatment, Session 1 will focus on psychoeducation, sessions 2-10 on ERP, 11-12 on relapse prevention.

All patients will voluntarily participate in assessments with the researcher while also completing self-reported measures. All clinician-rated assessments will be conducted with an independent evaluator (IE). The demographic data will be collected at the beginning of treatment, Baseline. The Y-BOCS and self-report Y-BOCS will be administered at Baseline and Post-treatment. The Clinical Global Impression-Severity, OCD Identity Questionnaire, Sheehan Disability Scale, Depression Anxiety Stress Scale-21 (DASS-21) Item Version and the Quality of Life (Q-LESQ-SF)-21 will be administered at Baseline, Mid treatment and Post-treatment to track patient symptomology. The weekly feedback measure will be administered every session to participants to collect data on their thoughts of how treatment is going. The following list of measures will be administered.

Researcher Administered:

1. Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
2. Self-report Yale-Brown Obsessive-Compulsive Scale
3. NIMH Global Obsessive-Compulsive Scale (NIMH-GOCS)
4. Clinical Global Impression-Severity/Improvement *

Self-Administered:

1. Demographic Form - Baseline
2. Sheehan Disability Scale- Baseline, Mid treatment and Post-treatment
3. OCD Identity Questionnaire- Baseline, Mid treatment and Post-treatment
4. Depression Anxiety Stress Scale - 21 Item Version (DASS-21) - Baseline, Mid treatment and Post-treatment
5. Quality of Life-21 (Q-LESQ-SF) - Baseline, Mid treatment and Post-treatment
6. Weekly Feedback Measure - Every session

The investigators will enroll all eligible subjects. A total of 70 individuals will participate. This number is anticipated based on group and individual dyad enrollment.

Descriptive analyses of participant data will be ongoing for one year, the entire duration of the study. For this study, descriptive statistics and symptomology improvements/ regressions analyses will be used to analyze study variables. Measures will be analyzed for use of future publications surrounding ERP treatment for OCD in groups and individual settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults 18 years or older.
* Participants must have the capacity and ability to give informed consent.
* Participants have been given an assessment and received a diagnosis of OCD.
* Participants must speak English.
* Participants must be able to physically attend treatment.

Exclusion Criteria:

* Prisoners or any other high-risk population group.
* experiencing active psychosis
* experiencing active substance abuse disorder
* experiencing active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale | Post-treatment, 6 weeks after baseline
  Participant OCD severity is measured with Yale-Brown Obsessive-Compulsive Scale over the course of their time in the study. Severity is measured at baseline (week 1), mid (week 3), and post (week 6) participation in ERP over the course of 6 weeks. Severity on the scale is measured based on a score range of 0-40. Participants with scores of 0-13 are considered to have mild symptoms. Scores of 14-25 are considered moderate. 26-34 are considered to be moderate-severe. 35-40 are considered to be very severe.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McIngvale, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine Jamail Building, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No